CLINICAL TRIAL: NCT02477579
Title: A Prospective, Multi-Center, Non-randomized, Single Arm, Open Label, Pivotal Study to Evaluate the Safety and Effectiveness of the NovaCross™ Micro-catheter in Facilitating Crossing Chronic Total Occlusion (CTO) Coronary Lesions
Brief Title: A Prospective, Multi-Center, Pivotal Study to Evaluate the Safety and Effectiveness of the NovaCross™ Micro-catheter in Facilitating Crossing Chronic Total Occlusion (CTO) Coronary Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nitiloop Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-CLP-01
Record Dates: First submitted 2015-06-17; First posted 2015-06-23 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Chronic Total Occlusion of Coronary Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NovaCross (Experimental): NovaCross microcatheter will be used.
  Interventions: Device: NovaCross

INTERVENTIONS:
Device: NovaCross — The NovaCross™ is a guidewire positioning and support microcatheter for improving chronic total occlusion (CTO) crossability. The NovaCross™ gains its supportive characteristics through the use of a unique operator-controlled Nitinol scaffold and an extendable segment, both at its distal tip.

SUMMARY:
This study evaluates the safety and effectiveness of the a novel device called NovaCross to help cross Chronic Total Occlusion (CTO) lesions in coronary arteries.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the safety and effectiveness of the NovaCross™ micro-catheter when used to facilitate crossing of Chronic Total Occlusion (CTO) lesions in coronary arteries. The procedure will be conducted on consenting patients diagnosed with a CTO in a coronary vessel that requires revascularization after a previously failed attempt to cross or refractory to 10 minutes of conventional guidewire attempt.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 25-80
* Patient understands and has signed the study informed consent form.
* Patient has an angiographic documented Chronic Total Occlusion (i.e. >3 months occlusion duration) showing distal TIMI flow 0.
* Suitable candidate for non-emergent, coronary angioplasty
* Documented coronary angiography preceding the PCI reveals at least one CTO lesion situated in a non-infarct related coronary artery or its side branches
* Body Mass Index (BMI) < 40
* Left ventricle ejection fraction > 25%

Exclusion Criteria:

* Patient unable to give informed consent.
* Current participation in another study with any investigational drug or device.
* Patient is known or suspected not to tolerate the contrast agent.
* Aorta-ostial CTO location (Ostial bifurcation origins may be considered), SVG CTO, in-stent CTO.
* Intolerance to Aspirin and/or inability to tolerate a second antiplatelet agent (Clopidogrel and Prasugrel and Ticagrelor).
* Appearance of a fresh thrombus or intraluminal filling defects.
* Recent major cerebrovascular event (history of stroke or TIA within 1 month)
* Cardiac intervention within 4 weeks of the procedure
* Renal insufficiency (serum creatinine of > 2.3mg/dl or 203μmol/L)
* Active gastrointestinal bleeding
* Active infection or fever that may be due to infection
* Life expectancy < 2 years due to other illnesses
* Significant anemia (hemoglobin < 8.0 mg / dl)
* Severe uncontrolled systemic hypertension (> 240 mmHg within 1 month of procedure)
* Severe electrolyte imbalance
* Congestive heart failure [New York Heart Association (NYHA) Class III\IV] CSA Class IV.
* Unstable angina requiring emergent percutaneous trans-luminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG)
* Recent myocardial infarction (MI) (within the past two weeks)
* Uncontrolled diabetes >2 serum glucose concentrations of >350 mg/dl within 7 days.
* Unwillingness or inability to comply with any protocol requirements
* Pregnant or nursing
* Extensive prior dissection from a coronary guidewire use
* Drug abuse or alcoholism.
* Patients under custodial care.
* Bleeding diathesis or coagulation disorder;
* Kawasaki's disease or other vasculitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-05-17 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
MACE | 30 days
  30 day MACE, defined as the composite of death, myocardial infarction (MI), or urgent revascularization (target vessel revascularization (TVR) or urgent coronary artery bypass surgery (CABG)).
Intra-procedural technical success | Intra-procedure
  Intra-procedural technical success, defined as the ability of the NovaCross™ micro-catheter to successfully facilitate placement of a guidewire beyond a native coronary chronic total occlusion (CTO) in the true vessel lumen.

SECONDARY OUTCOMES:
1. The ability to cross the lesion with a guidewire in the true lumen, effectively dilate the CTO lesion, and place a coronary stent with residual lumen stenosis of less than 30% while restoring antegrade TIMI 3 flow. | Procedure
  1. The ability to cross the lesion with a guidewire in the true lumen, effectively dilate the CTO lesion, and place a coronary stent with residual lumen stenosis of less than 30% while restoring antegrade TIMI 3 flow.
Proximal cap (ability of the NovaCross™ micro-catheter to facilitate a guidewire successfully penetrating the proximal cap of the CTO.) | Procedure
  2. The ability of the NovaCross™ micro-catheter to facilitate a guidewire successfully penetrating the proximal cap of the CTO.
Effectiveness of extendable portion (effectiveness of the extendable portion in intra-CTO microcatheter crossability) | Procedure
  3. The effectiveness of the extendable portion in intra-CTO microcatheter crossability.
Visualization (ability to have full visualization of the NovaCross during the CTO procedure) | Procedure
  4. The ability to have full visualization of the NovaCross during the CTO procedure.
Usability (Assess the usability of the NovaCross™ by the operator) | Procedure
  5. Assess the usability of the NovaCross™ by the operator.
Device-related perforation (at the site of target coronary lesion and/or its proximal reference segment) | Procedure
  6. Device-related perforation at the site of target coronary lesion and/or its proximal reference segment.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Walsh, MD, Principal Investigator — Belfast Health and Social Care Trust
Locations (5):
- United States (4):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Edward Hospital, Naperville, Illinois
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - York Hospital, York, Pennsylvania
- SPZOZ University Hospital in Krakow, Krakow, Poland